CLINICAL TRIAL: NCT03931967
Title: Proadrenomedullin and Microcirculation in Monitoring Organ Dysfunction in Patient With Infection: Prospective Observational Study
Brief Title: Proadrenomedullin and Microcirculation in Monitoring Organ Dysfunction in Patient With Infection
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Clinical Professor, Università Politecnica delle Marche
Other Study IDs: MicroMRproADM
Record Dates: First submitted 2019-03-05; First posted 2019-04-30 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-04

CONDITIONS: Infection; Sepsis; Septic Shock
Keywords: Sepsis; Septic shock; Microcirculation; Glycocalix; Proadrenomedullin; Organ dysfunction; Critical Care; Intensive Care
MeSH Terms: conditions — Infections; Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dosage of MicroMRproADM, endothelin-1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MR-proADM
  Interventions: Diagnostic Test: MR-proADM

INTERVENTIONS:
Diagnostic Test: MR-proADM — to evaluate the plasmatic level of MR-proADM and endothelin-1 in the first five days of ICU stay.

SUMMARY:
This study evaluates the association between plasmatic levels of Mid Regional Proadrenomedullin (MR-proADM) and the sublingual microcirculation in critical care patients admitted with infection, sepsis or septic shock.

DETAILED DESCRIPTION:
MR-proADM (Mid Region proAdrenomedullin) is a fragment of 48 amino-acids of ADM (Adrenomedullin), a protein belonging to the super-family of calcitonin-related peptides. MR-proADM is released in a 1:1 ratio with its native protein ADM. Blood levels of ADM are high in several conditions including infection, sepsis of septic shock. MR-proADM seems to be a promising marker for early diagnosis, prognosis and mortality in sepsis and it is also related to sepsis-induced organ failure.

The microcirculatory and endothelial damages represent two corner stones of the sepsis pathophysiology. They involved the loss of functional capillaries density and the loss of red blood cells deformability, the endothelial cell disfunction induced by sepsis, the induction of the apoptosis and necrosis, the alteration in the capillary permeability due to the loss of vasomotor tone and control. Moreover sepsis is characterised by the increased levels of adhesion molecules and the consequent interaction between neutrophils and endothelium, the fibrin deposition and the activation of the coagulation.

The aim of the study is to evaluate the correlation between the alteration in microcirculation and the levels of MR-proADM.

MFI (Microvascular Flow Index) is a qualitative measurement of microcirculation and the microcirculatory alterations during sepsis are crucial in the pathophysiology of this syndrome. It is related to prognosis and mortality in patient with sepsis in ICU (Intensive Care Unit)

Studying the relations between MFI and MR-proADM in the first five days of ICU stay could represent a good way to connect the pathophysiological background to a laboratory marker for an early diagnosis and for a measure of prognosis in patient with infections.

It is also important to compare the levels of MR-proADM with the other microcirculatory parameters (Total Vessel Density, Perfused Vessels Density, Percentage of Perfused Vessels, DeBacker score, Flow Heterogeneity index) and with the parameters of glycocalix and endothelial disfunction (Perfused Boundary Region and Endothelin-1)

When inclusion criteria are present and there are no exclusion criteria, patients will be enrolled for this five-days long study. Informed consent will be taken from the patient before enrollment or from the legal representative but when the neurological conditions do not allow

At the beginning of the study anthropometric data will be collected together with the main clinical and laboratory parameters (systolic, diastolic and mean arterial pressure, heart rate, mechanical ventilation parameters, blood gas parameters, vasoactive therapy, main parameters for renal, hepatic and haematological function, infectious condition and cultures).

Arterial blood samples will be collected and blood will be immediately centrifuged and plasma and serum samples will be stored at -80°C for the measurement of MR-proADM and Endothelin-1.

Moreover at the beginning of the study, the day after and the fifth days from the enrolment, the main microcirculatory parameters will be taken through Incident Dark Field Technology. Glycocheck Technology will be used to collect glycocalix conditions.

ELIGIBILITY:
Inclusion Criteria:

* Suspected Infection, Infection, Sepsis or Septic Shock in patient admitted in ICU from no more than 24 hours and which have previously monitored blood pressure and have a central venous catheter in place.

Exclusion Criteria:

* Age < 18 yo
* Length of stay in ICU > 24 hours;
* Length of stay in other hospital unit, ward or surgery > 48 hours;
* Refusal of informed consent;
* Conditions that do not allow the possibility of getting a monitoring of sublingual microcirculation (maxillofacial trauma, serious inability to jaw, copious blood loss or secretions from the mouth)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients with suspected infection, infection, sepsis or septic shock admitted to ICU
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Assessment of Microvascular Flow Index (MFI) | Five days
  Correlation between plasmatic value of MR-proADM and variation in Microvascular Flow Index (MFI) in patients admitted in ICU with suspected infection. MFI is detected in vivo by Incident Dark Field (IDF) Imaging at sublingual microcirculation. It represents the quality of blood flow at microcirculatory level.
Assessment of the concentration of Mid Regional Proadrenomedullin (MR-proADM) | Five days
  Correlation between plasmatic value of MR-proADM and variation in Microvascular Flow Index (MFI) in patients admitted in ICU with suspected infection. Mid Regional Proadrenomedullin (MR-proADM, unity of measurement nmol/L) is measured through a specify immunoenzymatic assay. MR-proADM is a diagnostic and prognostic marker of infection and sepsis.

SECONDARY OUTCOMES:
Cut-off for Microvascular Flow Index (MFI) based on Mid Regional Proadrenomedullin (MR-proADM) levels | Five days
  Founding a MR-proADM cut-off which would be able to predict a variation in MFI in patients admitted in ICU with suspected infection.
Assessment of patient's mortality | Five days
  Correlation between mortality (in percentage) and plasmatic levels of MR-proADM, based on MR-proADM clearance.
Assessment of new organ failure | Five days
  Correlation between organ failures and MRproADM, based on daily calculation of Sequential Organ Failure Assessment Score(SOFA score, 0 best value up to 24 worst value).Score subscales:Respiratory(PaO2/FiO2 (mmHg)≥ 400,score 0,< 400,+1,< 300, +2,< 200 and mechanically ventilated,+3,< 100 and mechanically ventilated,+4);Nervous(Glasgow coma scale 15,score 0,13-14,+1,10-12 +2,6-9 and mechanically ventilated,score +3,<6,+4);Cardiovascular(Mean arterial pressure/vasopressors:MAP≥70 mmHg,score 0,MAP<70 mmHg,+1,dopamine≤5 µg/kg/min or dobutamine (any dose),+2,dopamine>5 µg/kg/min OR epinephrine≤0.1 µg/kg/min OR norepinephrine≤ 0.1µg/kg/min,+3,dopamine>15 µg/kg/min OR epinephrine>0.1µg/kg/min OR norepinephrine>0.1µg/kg,+4);Liver(Bilirubin(mg/dl)[μmol/L],< 1.2[< 20],score 0,1.2-1.9[20-32],+1,2.0-5.9[33-101], +2,6.0-11.9[102-204],+3,> 12.0[> 204],+4);Kidney(Creatinine (mg/dl)[μmol/L] < 1.2[< 110],score 0,1.2-1.9[110-170],+1,2.0-3.4[171-299],+2,3.5-4.9[300-440],+3,> 5.0[> 440], +4),Coagulation
Assessment of Procalcitonine (PCT) | Five days
  Correlation between PCT (Unity of measurement, ng/ml) and MR-proADM as combined score for outcome measurement in term of mortality.
Assessment of other microcirculatory parameters in patient with sepsis or septic shock. | Five days
  Correlation between plasmatic value of MR-proADM and variation in Perfused Vessels Density (PVD, unity of measure 1/mm), Percentage of Perfused Vessels (PPV, unity of measure %), Total Vessels Density (TVD, unity of measure mm/mm2), Flow Heterogeneity Index (FHI), DeBacker Score (unit of measure, 1/mm). The parameters are detected in vivo by Incident Dark Field (IDF) Imaging at sublingual microcirculation. MR-proADM is a diagnostic and prognostic marker of infection and sepsis.
Mid Regional Proadrenomedullin (MR-proADM) in patient with difference infectious condition. | Five days
  Comparison of the MR-proADM blood concentration (nmol/L) in patient with suspected infection, infection, sepsis and septic shock.
Correlation between Mid Regional Proadrenomedullin (MR-proADM) and glycocalix and endothelial damage. | Five days
  Association between plasmatic value of MR-proADM and variation in Perfused Boundary Region (PBR, the parameters is detected in vivo by Sidestream Dark Field (SDF) Imaging at sublingual microcirculation) and Endothelin-1. MR-proADM is a diagnostic and prognostic marker of infection and sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Abele Donati, MD, PhD, Principal Investigator — UNIVERSITA' POLITECNICA DELLE MARCHE
Locations (1):
- AOU Ospedali Riuniti Ancona - Università Politecnica delle Marche, Ancona, Italy